CLINICAL TRIAL: NCT05380388
Title: A Phase II Clinical Study to Assess the Safety, Immunogenicity, and Efficacy of Blood-stage Plasmodium Vivax Malaria Vaccine Candidate PvRII/Matrix-M in Healthy Thai Adults Living in Thailand
Brief Title: A Safety, Immunogenicity and Efficacy Study of PvRII/Matrix-M in Healthy Thai Adults Living in Thailand ( MIST3 )
Acronym: MIST3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MAL22004
Record Dates: First submitted 2022-04-13; First posted 2022-05-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Plasmodium Vivax Infection; Malaria Vaccine
MeSH Terms: interventions — Malaria Vaccines; Matrix-M

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Malaria Vaccine (Experimental): PvRII/Matrix-M month 0, month 1, month 6
  Interventions: Biological: Malaria Vaccine
- control (Other): HBV vaccine month 0, month 1, month 6
  Interventions: Biological: HBV vaccine

INTERVENTIONS:
Biological: Malaria Vaccine — blood stage Plasmodium vivax malaria vaccine
  Other Names: PvRII/Matrix-M
  Arms: Malaria Vaccine
Biological: HBV vaccine — HBV Vaccine
  Arms: control

SUMMARY:
This project is the third part of a 5-year research program entitled "Malaria Infection Studies in Thailand (MIST)" and known as MIST3. MIST3's primary objectives are to assess the safety of the PvRII/Matrix-M vaccine candidate in healthy adult Thai volunteers and to establish whether the PvRII/Matrix-M vaccine can demonstrate a reduced parasite multiplication rate in vaccinated volunteers compared to a controlled group (placebo vaccine) in a blood-stage controlled human malaria infection model. This study will recruit up to 36 eligible healthy volunteers aged 20-55 in Thailand at the Faculty of Tropical Medicine, Mahidol University. Eighteen volunteers will receive three doses of the PvRII/Matrix-M candidate vaccine, and 18 volunteers will receive three doses of the placebo vaccine. Safety and immunogenicity will be evaluated after each dose as per protocol. Approximately four weeks after receiving the third vaccination, 24 volunteers will undergo blood-stage CHMI with Plasmodium vivax. The volunteers will be monitored closely as in-patients in the Hospital for Tropical Diseases and treated according to the Research Proposal Submission Form.

This study is funded by the UK Wellcome Trust. The grant reference number are Oxford/MORU: 212336/Z/18/Z and 212336/Z/18/A, and Mahidol University: 212336/A/18/Z and 212336/A/18/A

DETAILED DESCRIPTION:
Summary of trial design: Phase II, double-blinded, randomized controlled trial with CHMI, designed to assess the safety, immunogenicity, and protective efficacy of PvRII/Matrix-M vaccine.

Overview: This is a randomized controlled single-centre Phase II P. vivax blood-stage CHMI trial to assess the safety, immunogenicity, and efficacy of the candidate malaria vaccine PvRII/Matrix-M.

Healthy Thai adults aged between 20 and 55 years will be recruited and randomized at the Faculty of Tropical Medicine, Mahidol University in Bangkok.

Vaccination group: Up to 18 healthy adults aged between 20 and 55 years will be recruited. These volunteers will receive three doses of the PvRII/Matrix-M vaccine intramuscularly at months 0, 1, and 6.

Approximately three to four weeks post-boost (3rd vaccination), 12 volunteers will undergo P. vivax blood-stage CHMI, induced by injection of P. vivax infected erythrocytes.

Control group: Up to 18 healthy adults aged between 20 and 55 years will be recruited. These volunteers will receive three doses of HBV vaccine intramuscularly at months 0, 1, and 6.

12 volunteers will undergo P. vivax blood-stage CHMI, induced by injection of P. vivax infected erythrocytes.

Volunteers will have blood taken at regular intervals following vaccination and in the post-CHMI period to assess the immune response to vaccination and subsequent challenge, as well as parasite growth dynamics and gametocytaemia.

Close monitoring will continue until volunteers meet the criteria for treatment or until 28 days after the challenge, when treatment will be started empirically.

Therapy will be with a standard course of chloroquine where not contraindicated. As infection will be induced via intravenous injection of blood-stage parasites, there will be no liver-stage infection and no hypnozoite formation, thereby eliminating the need for radical cure with primaquine therapy. Follow-up at the study site will be up to 1 year after antimalarial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Thai adults aged 20 to 55 years
2. Minimum educational level of high school or equivalent
3. Red blood cells positive for the Duffy antigen/chemokine receptor (DARC)
4. Women only: Must practice continuous effective contraception for the duration of the study period until 3 months post-challenge.
5. Agreement to refrain from blood donation during the study and for 1 year after the initiation of antimalarial treatment.
6. Willing to be admitted to the Hospital for Tropical Diseases for clinical monitoring as required by the protocol until antimalarial treatment is completed and their symptoms are settling, willing to take a curative antimalarial treatment following CHMI, and willing to reside in Bangkok and its vicinity for 2 months after malarial treatment initiation.
7. Able to read and write in Thai.
8. Provide written informed consent to participate in the trial
9. Answer all questions on the informed consent quiz correctly
10. Completed COVID-19 vaccination with 2 doses of any WHO-approved vaccine

Exclusion Criteria:

1. Positive malaria qPCR OR malaria film prior to vaccination and challenge
2. Presence of any medical condition (either physical or psychological) that, in the judgment of the investigator, would place the participant at undue risk (including the history of clinically significant contact dermatitis) or interfere with the results of the study (e.g., underlying cardiac, renal, hepatic or neurological disease; severe malnutrition; congenital defects or febrile condition)
3. Presence of chronic disease or chronic use of medication
4. Prior receipt of other investigational vaccine which is likely to impact the interpretation of the trial data as assessed by the Investigator.
5. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection, asplenia, history of splenectomy, recurrent severe infections, and chronic infection
6. Immunosuppressant medication within the past 6 months preceding enrolment (D0) or plan to use during the study (inhaled and topical steroids are allowed)
7. History of allergic disease or reactions likely to be exacerbated by malaria infection
8. Female participant who is pregnant as evidenced by positive beta-human chorionic gonadotropin (β-HCG) test, or who is lactating or planning pregnancy during the course of the study.
9. Contraindications to the use of antimalarial treatment (e.g., chloroquine, atovaquone/proguanil, or dihydroartemisinin/piperaquine)
10. Use of medications known to have potentially clinically significant interaction with the antimalarial drugs that will be used in this study (chloroquine, atovaquone/proguanil, or dihydroartemisinin/piperaquine)
11. History of cardiac arrhythmia, including clinically relevant bradycardia or Known existing positive family history in both 1st AND 2nd-degree relatives < 50 years old for cardiac disease
12. Family history of congenital QT prolongation or sudden death
13. Any clinical condition, including using medications known to prolong the QT interval or screening electrocardiogram (ECG), demonstrates a QTc interval ≥ 450 ms.
14. Suspected or known history of alcohol abuse or history of drug abuse.
15. Concurrently participating in another clinical study, at any time during the study period
16. Positive hepatitis B surface antigen or seropositive for hepatitis C virus, or HIV
17. Finding on safety laboratory values as defined below:

    * Abnormal ALT [>upper normal range]
    * Abnormal serum creatinine [>upper normal range]
    * Clinically significant abnormalities in corrected calcium and magnesium blood levels
    * Haemoglobin < 11 g/dL
18. Blood group Rhesus negative
19. Blood incompatibility to the inoculum
20. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
21. Any history of anaphylaxis in reaction to vaccinations

Vaccination and re-vaccination exclusion criteria

1. Acute disease at the time of vaccination. (acute disease is defined as the presence of a moderate or severe illness with or without fever).

The following adverse events associated with vaccine immunisation constitute absolute contraindications to further vaccine administration. If any of these events occur during the study, the participant must be withdrawn and followed until the resolution of the event, as with any adverse event:

1. Anaphylactic reaction following administration of the vaccine
2. Pregnancy

Exclusion criteria on the day of CHMI

The following constitute absolute contraindications to CHMI:

1. Acute disease, defined as a moderate or severe illness with or without fever
2. Pregnancy
3. Use of systemic antibiotics with known antimalarial activity in the 30 days before challenge (e.g., trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, and azithromycin)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
solicited local adverse event | 7 days following each vaccination
  occurrence of solicited local reactogenicity signs and symptoms
solicited systemic adverse event | 7 days following each vaccination
  occurrence of solicited systemic reactogenicity signs and symptoms
unsolicited adverse events | 28 days following each vaccination
  Occurrence of unsolicited adverse events
safety laboratory measures | 28 days following each vaccination
  Number of participants with abnormal laboratory test results
serious adverse events | through study completion, an average of 1 year
  Occurrence of serious adverse events during the whole study duration
feasibility of primary P. vivax blood-stage CHMI | within 21 days following CHMI
  successful infection (development of detectable persistent parasitaemia by thick blood film +/- clinical symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Day, MD, Principal Investigator — University of Oxford
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, suitably anonymised clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future.

DOCUMENTS (1):
  • Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT05380388/Prot_000.pdf